CLINICAL TRIAL: NCT04814667
Title: LAROTRACKING - A Retro-/Prospective, Non-interventional, Cohort Study in Adult Patients With Locally Advanced or Metastatic Tumors With a Neurotrophic Tyrosine Receptor Kinase (NTRK) Gene Fusion, Treated With Larotrectinib
Brief Title: A Retro-/Prospective, Non-interventional, Cohort Study in Adult Patients With Locally Advanced or Metastatic Tumors With a Neurotrophic Tyrosine Receptor Kinase (NTRK) Gene Fusion, Treated With Larotrectinib
Acronym: LAROTRACKING
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: LAROTRACKING
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumor, Adult; Locally Advanced Solid Tumor; Metastatic Cancer
Keywords: NTRK gene fusion; Larotrectinib; Neurotrophic Tyrosine Receptor Kinase gene fusion; NTRK rearrangements
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Larotrectinib, a selective TRK inhibitor has showed marked and durable antitumor activity in patients with NTRK gene-fusion-positive tumors regardless of the tumor type, gene partner and patient's age. Because of this and the lack of alternative therapy in this rare but severe disease, the French National Agency for Medicines and Health Products Safety (ANSM) granted in April 2019, a "cohort" Temporary Authorization for Use (ATU) in the indication:"Larotrectinib is indicated as monotherapy for the treatment of adult and paediatric patients from one month, with locally advanced or metastatic solid tumours with a Neurotrophic Tyrosine Receptor Kinase (NTRK) fusion, refractory to standard treatments or in the absence of appropriate therapeutic alternative." Despite the potential benefit of identifying these fusions, the clinicopathologic features of NTRK fusion-positive tumors which are treated with Larotrectinib, are not well characterized. This study will provide information about the diagnosis and management of patients with locally advanced or metastatic NTRK fusion cancer treated with Larotrectinib under real-world treatment conditions in France, and describes the dosing patterns, safety and effectiveness of this agent.

DETAILED DESCRIPTION:
Tropomyosin receptor kinases (TRK) are a family of tyrosine kinases that bind neurotrophins, a family of growth factors important to the formation and function of the nervous system. In cancer, the neurotrophic tyrosine kinase receptor (NTRK)1, NTRK2 and NTRK3 genes, which encode for the TRKA, TRKB and TRKC proteins, respectively, are subject to gene-arrangements that lead to kinase domain expression and constitutive downstream pathway activation. In preclinical models, NTRK gene fusions have transformative oncogenic potential, and they appear to be widely distributed across histologically diverse adult and pediatric cancers. Hence, these genetic abnormalities, observed in both children and adults, have recently emerged as targets for cancer therapy.

Larotrectinib, a selective TRK inhibitor has showed marked and durable antitumor activity in patients with NTRK gene-fusion-positive tumors regardless of the tumor type, gene partner and patient's age.

Because of this and the lack of alternative therapy in this rare but severe disease, the French National Agency for Medicines and Health Products Safety (ANSM) granted in April 2019, a "cohort" Temporary Authorization for Use (ATU) in the indication:

"Larotrectinib is indicated as monotherapy for the treatment of adult and paediatric patients from one month, with locally advanced or metastatic solid tumours with a Neurotrophic Tyrosine Receptor Kinase (NTRK) fusion, refractory to standard treatments or in the absence of appropriate therapeutic alternative." Despite the potential benefit of identifying these fusions, the clinicopathologic features of NTRK fusion-positive tumors which are treated with Larotrectinib, are not well characterized.

This study will provide information about the diagnosis and management of patients with locally advanced or metastatic NTRK fusion cancer treated with Larotrectinib under real-world treatment conditions in France, and describes the dosing patterns, safety and effectiveness of this agent.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients
* Histological confirmed diagnosis of advanced/metastatic solid tumor type.
* Patients previously, currently or to be treated with Larotrectinib within the ATU/post-ATU period. Patient must be > 25 years-old at time of larotrectinib start.
* Patients not opposed to collection of personal clinical data

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with locally advanced or metastatic tumors with a Neurotrophic Tyrosine Receptor Kinase (NTRK) gene fusion, treated with Larotrectinib
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Clinical activity of larotrectinib | From the date of the first larotrectinib dose until the date of objectively documented progression or date of subsequent anti-cancer therapy, whichever came first, assessed up to 60 months.
  Best objective response rate (BORR) (Complete Response or Partial Response according to RECIST V1.1 classification i.e assessed by investigators)
Clinical activity of larotrectinib | From the start of Complete Response or Partial Response (whichever response came first) until the date of observed disease progression or death due to any cause, whichever came first, assessed up to 60 months.
  Duration of response (DOR) (Best overall response of Complete Response or Partial Response according to RECIST V1.1 classification i.e assessed by investigators)
Clinical activity of larotrectinib | From the start of larotrectinib treatment until the first evidence of Objective Response according to RECIST V1.1 classification i.e assessed by investigators), assessed up to 60 months. Time to response will be calculated for responders only.
  Time to response (TTR)
Clinical activity of larotrectinib | From the start of Larotrectinib treatment until the date of first observed disease progression (radiological or clinical, whichever came first) or death due to any cause, whichever came first, assessed up to 60 months
  Progression-free survival (PFS)
Clinical activity of larotrectinib | From the start of larotrectinib treatment until the date of death, due to any reason, assessed up to 60 months. Patients alive or lost to follow-up at the time of analysis will be censored at their last date of follow-up.
  Overall survival (OS)

SECONDARY OUTCOMES:
Clinicopathological features of patients with locally advanced or metastatic NTRK fusion cancer for whom a decision to treat with larotrectinib was made before enrolment. | Through study completion, an average of 60 months.
  Demographics data, significant or relevant medical history, cancer disease overview
Diagnosis strategy for detection of NTRK fusions in the investigational centers | Through study completion, an average of 60 months.
  Description of the diagnosis tests used for NTRK fusions
Treatment(s) received prior to and after larotrectinib. | From the first dose of larotrectinib until the day of permanent discontinuation of larotrectinib (including death), assessed up to 60 months .
  Doses, duration, best tumor response and reasons for discontinuation
Patterns of larotrectinib treatment | From the start of larotrectinib treatment until the day of permanent discontinuation of larotrectinib (including death), assessed up to 60 months
  Dosing paramaters
Safety of larotrectinib | Through study completion, an average of 60 months.
  Adverse events : Nature, frequency and severity of Adverse Events (AEs), Serious Adverse Events (SAEs) and Suspected Unexpected Serious Adverse Reactions (SUSARs) graded using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
Molecular characteristics of NTRK rearrangements | Through study completion, an average of 60 months.
  Gene name, type of alteration

CONTACTS AND LOCATIONS:
Overall Officials: Armelle DUFRESNE, Principal Investigator — Centre Leon Berard
Locations (4):
- France (4):
  - CHU Amiens, Amiens
  - Centre Georges Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Chi Elbeuf Louviers, Saint-Aubin-lès-Elbeuf